CLINICAL TRIAL: NCT06899906
Title: Efficacy and Safety of Dalbavancin As Suppressive Therapy
Acronym: DALBA-SAT
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 25-5019
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Efficacy and Safety of Dalbavancin; In Subjects Who Received SAT with DAL; For Acute or Chronic Infections Between July 2019 and December 2024

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Dalbavancin (DAL) as suppressive therapy (SAT): The study population included subjects aged ≥ 18 years who received SAT with DAL for acute or chronic infections (defined as a long-standing infection due to a previously uneradicated pathogen, following unsuccessful antibiotic or surgical treatments) between July 2019 and December 2024.
  Subjects younger than 18 years and those who received DAL not for SAT purposes were excluded.
  Interventions: Other: Determine patient demographic and clinical characteristics at baseline

INTERVENTIONS:
Other: Determine patient demographic and clinical characteristics at baseline — Description of demographic data (sex, age), comorbidities (Charlson scores), septic history, and medical management (antibiotic therapy)

SUMMARY:
Dalbavancin (DAL) is a semi-synthetic antibiotic that belongs to the lipoglycopeptide family and is structurally derived from teicoplanin, respect of which it has two structural differences that enhance its anti-staphylococcal binding affinity and extend its half-life to between 149 and 250 hours. It achieves adequate tissue penetration in the skin, bones, joints, lung tissues, and peritoneal space, maintaining concentrations above the MIC for susceptible Gram-positive pathogen.

DAL is a bactericidal antimicrobial agent that binds the C-terminal D-alanyl-D-alanine on the bacterial cell wall, blocking trans-glycosylation and transpeptidation processes essential for cell wall synthesis. It seems also to be able to enhance neutrophil antibacterial activity improving PMNs' intracellular killing of MRSA. It has also a good antibiofilm activity, alone or in combination with other molecules. Like other glycopeptide molecules, DAL shares a similar spectrum of activity, with demonstrated in vitro activity against various Gram-positive bacteria, including Staphylococcus spp, Streptococcus spp and Enterococcus (faecium, and faecalis). Resistance to DAL is possible in these gram-positives bacteria, given to presence of enzymes that produce low-affinity binding precursors for the antibiotic's binding site. DAL is capable to overcome Van-B mechanism of resistance, but it results not active in producing Van-A strains.

The study objectives was to evaluate efficacy and safety of DAL treatment.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Patients received SAT with DAL for acute or chronic infections (defined as a long-standing infection due to a previously uneradicated pathogen, following unsuccessful antibiotic or surgical treatments) between July 2019 and December 2024
* Patient who was informed and did not object to participating in the study

Exclusion Criteria:

* -< 18 years
* Subjects who received DAL not for SAT purposes

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients managed for gram-positive infection between July 2019 and December 2024 in the MIT department.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of DAL treatment, measured as the proportion of stable infection | Outcome will be measure at 1 year. For patients lost of follow-up or followed-up less than a year, the date of last visit will be used for survival curve analysis .

CONTACTS AND LOCATIONS:
Locations (1):
- HCL, France, Lyon, France